CLINICAL TRIAL: NCT06987435
Title: Investigation of the Flexibility of Structures Around the Ankle in Individuals With Chronic Ankle Instability
Brief Title: Elasticity of Structures Around the Ankle in Chronic Ankle Instability
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Busra Seckinogullari Korkusuz, Principal Investigator, Hacettepe University
Other Study IDs: 604.01.02-423
Record Dates: First submitted 2025-05-16; First posted 2025-05-23 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-05

CONDITIONS: Chronic Ankle Instability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to examine the flexibility of the structures around the ankle in individuals with unilateral chronic ankle instability. Individuals between the ages of 18-45 who have been diagnosed with chronic ankle instability by an orthopedist and who have unilateral instability will be included in the study. The flexibility of the healthy and instability sides will be evaluated. Demographic information of the individuals will be recorded and clinical evaluations will be made. The severity of ankle instability will be evaluated with the Functional Ankle Identification (FABIT). The foot posture of the individuals participating in the study will be evaluated with the Foot Posture Index, and the degree of flat feet will be evaluated with the Navicular Drop Test. The flexibility of the gastrocnemius, tibialis anterior, peroneus longus, achilles tendon and plantar fascia of the individuals participating in the study will be measured with a myotonometer.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 45
* Mini Mental State Exam (MMSE) score of 24 to 30
* Diagnosed with unilateral chronic ankle instability by a physician

Exclusion Criteria:

* Inability to communicate verbally
* Use of a walking aid
* Any history of lower extremity surgery
* People with severe visual impairment, neurological disorders and/or congestive heart failure.

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: Individuals with Chronic Ankle Instability
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Functional Ankle Identification | Baseline
  The Functional Ankle Identification method is a scale developed to evaluate the functional ankle instability of individuals.
Foot Posture Index | Baseline
  Foot Posture Index will be applied in this study to evaluate the foot postures of the participants.
Navicular Drop Test | Baseline
  The Navicular Drop Test will be administered to measure how much the participants' navicular bones have fallen.
Myoton | Baseline
  Participants' gastrocnemius, tibialis anterior, peroneus longus, achilles tendon and plantar fascia flexibility will be evaluated using a myotonometer device.

CONTACTS AND LOCATIONS:
Overall Officials: Süleyman Korkusuz, PhD, Study Chair — Atılım University; Büşra Seçkinoğulları Korkusuz, PhD, Principal Investigator — Ankara University
Locations (1):
- Atılım University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tas S, Salkin Y. An investigation of the sex-related differences in the stiffness of the Achilles tendon and gastrocnemius muscle: Inter-observer reliability and inter-day repeatability and the effect of ankle joint motion. Foot (Edinb). 2019 Dec;41:44-50. doi: 10.1016/j.foot.2019.09.003. Epub 2019 Sep 29. PMID 31704588
- [Background] Rydahl SJ, Brouwer BJ. Ankle stiffness and tissue compliance in stroke survivors: a validation of Myotonometer measurements. Arch Phys Med Rehabil. 2004 Oct;85(10):1631-7. doi: 10.1016/j.apmr.2004.01.026. PMID 15468023
- [Background] Redmond AC, Crosbie J, Ouvrier RA. Development and validation of a novel rating system for scoring standing foot posture: the Foot Posture Index. Clin Biomech (Bristol). 2006 Jan;21(1):89-98. doi: 10.1016/j.clinbiomech.2005.08.002. Epub 2005 Sep 21. PMID 16182419